CLINICAL TRIAL: NCT00328809
Title: Subjects With Severe Heart Failure and End-Stage Renal Disease on Hemodialysis: A Pilot Study to Assess Safety and Tolerability of Spironolactone
Brief Title: Spironolactone Safety in Dialysis Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: personnel shortage
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, Sri Narsipur, Associate Professor of Medicine and Pediatrics, State University of New York - Upstate Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1045057
Record Dates: First submitted 2006-05-19; First posted 2006-05-22 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: End Stage Renal Disease; Congestive Heart Failure
MeSH Terms: conditions — Kidney Failure, Chronic; Heart Failure | interventions — Spironolactone

ARMS (1):
- Spirnolactone (Experimental)
  Interventions: Drug: spironolactone

INTERVENTIONS:
Drug: spironolactone — spironolactone administered to ESRD patients at low dose

SUMMARY:
Cardiovascular disease is the leading cause of death and disproportionately prevalent in patients with kidney disease. Spironolactone has been shown to improve survival in the general population with heart failure by up to 30%. We wish to study the safety and tolerability of aldosterone blockade with spironolactone on cardiac function in a high risk population of patients on hemodialysis. We will study and closely monitor subjects over a period of 12 months, during which they will be receiving spironolactone for a period of 6 months.

ELIGIBILITY:
Inclusion Criteria:

* They must be at least 18 years of age.
* They must understand the study purpose and give their written informed consent.
* They must have been stable on chronic hemodialysis for at least three months before enrollment into the study.
* Hemodialysis subjects will be included if they have had a left ventricular ejection fraction measured within the past six months with a value no more than 45 percent. A repeat, standardized echocardiogram will be used to confirm left ventricular ejection fraction.

Exclusion Criteria:

* Subjects with primary operable valvular heart disease.
* Subjects with a congenital heart disease.
* Subjects with unstable angina.
* Subjects with primary hepatic failure.
* Subjects with active cancer or any life-threatening disease (other than heart failure or end-stage renal disease).
* Subjects who have undergone heart transplantation or who are awaiting heart transplantation are also ineligible.
* Subjects on a renal transplant list will be accepted into the study until the time of successful renal transplantation and termination of dialysis.
* Subjects with habitually difficult to control hyperkalemia (serum potassium >6.0 meq/L) in the previous month while on dialysis will be excluded.
* The inability to complete the 6-minute walk test will not be a reason to exclude subjects from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-06-30 (Estimated); Primary Completion 2017-06-30 (Estimated); Study Completion 2019-09-24 (Actual)

PRIMARY OUTCOMES:
risk of hyperkalemia | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sriram S Narsipur, MD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States

REFERENCES:
- [Derived] Hasegawa T, Nishiwaki H, Ota E, Levack WM, Noma H. Aldosterone antagonists for people with chronic kidney disease requiring dialysis. Cochrane Database Syst Rev. 2021 Feb 15;2(2):CD013109. doi: 10.1002/14651858.CD013109.pub2. PMID 33586138